CLINICAL TRIAL: NCT06828588
Title: Pilot Study of [68Ga]Ga-ABY-025 Imaging in Patients Undergoing Treatment With HER2-targeted Therapy
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, Eben Rosenthal, Barry and Amy Baker Professor and Chair, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VICCBREP24601
Record Dates: First submitted 2025-01-29; First posted 2025-02-14 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Cancer; Metastatic Cancer; HER2; HER2 + Breast Cancer, HER2 + Gastric Cancer, Squamous Cell Carcinoma of Head and Neck, Esophageal Squamous Cell Carcinoma; HER 2 Low-expressing Breast Cancer
Keywords: HER2; cancer; advanced cancer; metastatic; IHC; FISH; trastuzumab; T-DM1; Pertuzumab; Margetuximab; Neratinib; Lapatinib; Tucatinib; Everolimus
MeSH Terms: conditions — Neoplasm Metastasis; Breast Neoplasms; Stomach Neoplasms; Esophageal Squamous Cell Carcinoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study Arm (ABY-025) (Experimental): This is a pilot study of [68Ga]Ga-ABY-025, a radiolabeled affibody, imaging in patients undergoing treatment with HER2-targeted therapy. The PET/CT imaging ("HER2 PET" imaging) will be performed at, prior to, or during the time a patient is receiving treatment with HER2-targeted therapy. A second HER2 PET will be collected at time of therapy treatment discontinuation or 12 months from study consent. Patients will be infused with the study drug, Ga-ABY-025, on Day 0, followed by PET/CT imaging post infusion. Participants will undergo follow-up visits to assess for adverse reactions at 24 hours and 21 days post infusion (± 7 days). Participants will undergo standard of care work-up for their malignancy as determined by their treatment team (e.g. biopsy, additional imaging, observation, treatment for metastatic disease). Either at 12 months after enrollment in the study or at the time of treatment discontinuation (whichever comes first), repeat HER2 PET imaging will
  Interventions: Drug: ABY-025 Loading Dose; Drug: [68Ga]Ga-ABY-025

INTERVENTIONS:
Drug: ABY-025 Loading Dose — Subjects will receive a loading dose (400 micrograms) of ABY-025 prior to the [68Ga]Ga-ABY-025 infusion.
Drug: [68Ga]Ga-ABY-025 — Subjects receive a tracer dose of [68Ga]Ga-ABY-025 and will receive a PET/CT scan a few hours after the injection.

SUMMARY:
The purpose of this study is to determine if the radiotracer, [68Ga]Ga-ABY-025, used for PET imaging can help us better identify and visualize lesions or tumors, in patients who are receiving standard of care therapy HER2+ cancers.

DETAILED DESCRIPTION:
This study will assess a dose of ABY-025 followed by a tracer dose of [68Ga]Ga-ABY-025 in subjects with HER2+ solid cancers, or HER2+ or low breast cancer undergoing or planning to undergo treatment with standard-of-care HER2-targeted therapy for an FDA-approved indication. The study drug will be administered on Day 0, and [68Ga]Ga-ABY-025 PET/CT scan will be obtained the same day after injection of study drug. Patients will receive a phone call from a study coordinator post-injection to assess for adverse events. Subjects will undergo standard of care evaluation of their advanced disease per the discretion of their treating physician.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Patients with unresectable locally advanced or metastatic cancer who are eligible for standard of care treatment with HER2-targeted therapy per the discretion of their treating physician for an FDA-approved indication. Patients who are planning to start HER2-targeted therapy at the time of study enrollment. Patients who have recently begun HER2 treatment and have received no more than 6 cycles will be eligible for enrollment.
3. Must have a previous biopsy demonstrating HER2 expression in at least one lesion (HER2+ solid cancer, or breast cancer patients who are HER2+ or HER2-low) as defined by IHC and FISH studies or with HER2 amplification as defined by a liquid biopsy that was done as standard of care testing for the patient's cancer type.
4. Measurable disease on CT, FDG-PET, or MRI imaging for RECIST evaluation; patient must have measurable disease outside the liver.
5. Life expectancy of at least 6 months. Patients with brain metastases are permitted to enroll in this study.

Exclusion Criteria:

1. Measurable sites of disease only in the liver.
2. Inability to comply with study procedures.
3. Hypersensitivity or allergy to any component of [68Ga]Ga-ABY-025.
4. Pregnant or breastfeeding.
5. HER2-negative cancers that have no FDA approved indication for treatment with HER2-directed therapy.
6. Inability to lie flat for 30 minutes during an imaging session.
7. Medical or psychiatric co-morbidities that, in the opinion of the treating physician, would prevent the patient from successfully participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Determine safety of [68Ga]Ga-ABY-025 PET by assessing for adverse events following the injection and PET imaging. | up to 21± 14 days from second administration of [68Ga]Ga-ABY-025. Assessments will be performed as part of the routine standard of care for patients undergoing HER2-targeted anti-cancer treatment.
  Outcome Measure: After study enrollment, subjects will receive [68Ga]Ga-ABY-025 infusion and undergo PET/CT scan. Patients will be immediately assessed for adverse events within the first 30 minutes of infusion and via phone call at 2 days (± 1 day) post-infusion from the study coordinator. Adverse events will be monitored up to 21±14 days following the infusion of study drug. Repeat infusion and imaging will be obtained either at the time of treatment discontinuation or at 12 months from study consent and will have the same safety monitoring parameters. While there are expected adverse events related to anti-cancer therapy, we will specifically be reporting adverse events that are "definitely related" or "probably related" to the study agent.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is unknown if and/or how we will plan IPD with outside researchers.

DOCUMENTS (1):
  • Informed Consent Form (2025-04-16): https://cdn.clinicaltrials.gov/large-docs/88/NCT06828588/ICF_000.pdf